CLINICAL TRIAL: NCT03848702
Title: Nonoperative Treatment of Dorsally Dislocated Distal Radius Fractures in Adults With an Individualized 3D Printed Brace; a Tolerability Study in Healthy Volunteers and Patients (DRFB)
Brief Title: Nonoperative Treatment of Dorsally Dislocated Distal Radius Fractures in Adults With an Individualized 3D Printed Brace.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VieCuri Medical Centre (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Nl61002.078.17
Record Dates: First submitted 2019-02-13; First posted 2019-02-21 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Dorsal Displacement

STUDY DESIGN:
Intervention Model Description: Two consecutive prospective case series to investigate brace feasibility.
Who Masked: Participant, Care Provider
Masking Description: For part 1, a randomization list will be generated using an online program. For the 10 participants, five braces will be developed for the dominant side and five for the nondominant side. The physician and participant will be concealed for allocated side until the scan will be made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Experimental): All volunteers wore the DRFB
  Interventions: Device: Distal radius fracture brace
- Patients with DRF (Experimental): All patients wore the DRFB
  Interventions: Device: Distal radius fracture brace

INTERVENTIONS:
Device: Distal radius fracture brace — The distal radius fracture brace is constructed from biocompatible materials (like polylactic acid; PLA) and the skin is protected by commercially available and approved waterproof padding (like Aquacast®). The major brace components are connected and reinforced with carbon rods and plastic bolt-nut connections. PLA is extensively used, for example in surgical implants, but also as biological alternative for plastics. Aquacast® is approved and used as waterproof padding in swim plaster. The biomechanical function of the distal radius brace has been tested successfully in an ex vivo setting (results to be published). The DRFB includes the distal forearm, wrist an base of the hand. The thumb and fingers are free and the DRFB provides more movement than classical casting.

SUMMARY:
Study design: Two consecutive prospective case series. Study population: Part 1 will enroll 10 healthy volunteers (50 years or older). Part 2 will enroll 10 elderly patients (50 years or older) with a dorsally displaced distal radius fracture (AO type 23-A-C) that is acceptably reduced. In both parts, participants should have no restrictions in activities of daily living pre-fracture and no evident anatomical difference between both wrists.

Intervention:

Part 1: Participants will wear the brace continuously for one week. Part 2: Participants will wear the brace as treatment of the fracture for five weeks (instead of a plaster cast).

Main study parameters/endpoints: In parts 1 and 2, the primary outcome measure will be a Visual Analog Scale (VAS) score for wearing comfort. Secondary outcome measures are the occurrence of fracture redislocation (part 2 only), pain (VAS), inconvenience during NL61002.078.17 / DRFB-Tolerability Distal Radius Fracture Brace Tolerability Version number: 1.1, d.d. April 24, 2017 8 of 34 activities of daily living (Katz Index), and adverse reactions like pain, skin pressure, skin irritation/redness, sensibility issues, or device-related problems.

DETAILED DESCRIPTION:
Rationale: Each year, approximately 34,500 adults in The Netherlands sustain a fracture of the distal radius (wrist fracture). Incidence peaks in the elderly. The currently preferred treatment is closed reduction and nonoperative treatment by immobilization in a plaster cast for 4-6 weeks. Surgery is only performed if closed reduction fails or redislocation occurs. Plaster immobilization is inconvenient and interferes with daily activities. More importantly, standard nonoperative treatment often fails; in 40-60% of the fractures, redislocation requires surgery. Surgical treatment is about 9 times more expensive than nonoperative treatment and not without risks. This project aims to develop an innovative nonoperative treatment option. The central idea is to produce a 3D-printed brace for the fractured wrist using a mirrored CT-scan of the contralateral, unfractured wrist as a model. This innovative approach has the advantage that it does not depend on surgery and provides a better and potentially more durable positioning than the currently applied plaster cast. We expect that redislocation will occur less frequently, so surgery may be avoided. In contrast to a traditional plaster cast, the newly developed brace is water resistant/repellant, lighter, and enables movement of the hand. It enables daily activities and improves independency in the elderly with a wrist fracture. The treatment has been successfully evaluated in an ex vivo model. The clinical implementation will follow a step-wise approach.

Objective: Part 1 aims to determine the tolerability of the 3D-printed brace when worn by healthy volunteers (50 years of order), performing their normal daily activities. In part 2, the objective is to determine tolerability of the 3D-printed brace in patients (50 years or older) with an extra-articular distal radius fracture with dorsal displacement, performing their normal daily activities.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

1. Age 50 years or older
2. Healthy volunteer without distal radius fracture
3. No restrictions in activities of daily living prior to enrolment*
4. Signed informed consent by participant * Participant should exercises complete self-control over urination and defecation, but use of incontinence material is allowed.

Part 2:

1. Patients (50 years or older) with an acute**, unilateral distal radius fracture with dorsal displacement (AO type 23-A, B, or C) that is acceptably reduced (by simple closed reduction with vertical longitudinal traction)
2. No restrictions in activities of daily living pre-fracture*
3. Signed informed consent by patient

   * Participant should exercises complete self-control over urination and defecation, but use of incontinence material is allowed. ** Patients should report to the Emergency Department within 48h post-trauma.

Exclusion Criteria:

Part 1:

1. Preexisting anatomical deviation of the ipsi- or contralateral wrist
2. Conditions that affect function of the wrist or hand
3. Insufficient comprehension of the Dutch or language to understand the study documents
4. Participant unwilling or unable to comply with the study protocol and follow-up visit schedule
5. Known allergy for brace material (PLA or alternative)

Part 2:

1. Preexisting anatomical deviation of the ipsi- or contralateral wrist
2. Additional traumatic injuries that affect treatment, rehabilitation, or function of the affected hand
3. Pathological, recurrent, or open fracture
4. Impaired wrist function pre-trauma at either wrist (e.g., arthrosis, rheumatoid disorder, or neurological disorder)
5. Bone disorder that may impair bone healing, excluding osteoporosis
6. Patient unwilling or unable to comply with the treatment protocol and follow-up visit schedule
7. Insufficient comprehension of the Dutch language to understand the study documents
8. Known allergy for brace material (PLA or alternative).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
VAS score | Day 1, day 3 and 7 for part 1. Week 1, week 2 and week 5 for part 2
  the primary outcome measure will be the change in 1 week (part 1) and over several weeks (part 2) on a 10-centimeter Visual Analog Scale (VAS) score for wearing comfort, in which 0 implies no comfort. and 10 implies extremely comfortable.

SECONDARY OUTCOMES:
Redislocation | Week 1, week 2 and week 5 (only part 2)
  Redislocation is determined by the radiologic outcome:
  * Dorsal tilt > 15˚ on lateral X-ray
  * Volar tilt >20˚ on lateral X-ray
  * Shortening >5mm pertaining to the ulna in PA direction
  * Intraarticular step-off ≥ 2mm
  * Radial inclination < 15˚ in PA direction
  * Subluxation of the lunate According to guidelines on these parameters, redislocation is diagnosed.
Pain Level | Day 1, day 3 and 7 for part 1. Week 1, week 2 and week 5 for part 2
  Pain level caused by the brace will be determined using a 10-centimeter Visual Analog Scale (VAS), in which 0 implies no pain and 10 implies the worst possible pain.
Inconvenience | Day 1, day 3 and 7 for part 1. Week 1, week 2 and week 5 for part 2
  Inconvenience during activities of daily living using the Katz Index. The Katz Index asks for limitations in washing, clothing, indoor transfers, toilet visit, continence and eating. The range for the Katz index is 0 to 6 where 6 indicates full function, 4 indicates moderate impairment and 2 or less indicates severe functional impairment.
Adverse reactions (pain, skin pressure, skin irritation/redness, sensibility issues or device-related problems | Day 1, day 3 and 7 for part 1. Week 1, week 2 and week 5 for part 2
  Adverse reactions like pain, skin pressure, skin irritation/redness, sensibility issues, or device-related problems.

OTHER OUTCOMES:
Age (calculated from date of birth and date of enrolment) | At baseline
  - Age (calculated from date of birth and date of enrolment)
Gender | At baseline
  - Gender (male or female)
ASA class | At baseline
  - ASA class (1, 2, 3 of 4), assessed in a face-to-face interview
BMI (calculated from height and weight) | At baseline
  - BMI (calculated from height and weight)
Tobacco consumption | At baseline
  - Tobacco consumption (current, ever, never) was assessed in a short face-to-face interview
Alcohol consumption | At baseline
  - Alcohol consumption at enrolment (yes or no), assessed in a face-to-face interview
Comorbidities including osteoporosis | At baseline
  - Comorbidities including osteoporosis were assessed from the electronic patients dossiers
Medication use | At baseline
  Medication use was assessed through the electronic patient dossiers
Dominant side (left or right) | At baseline
  Dominant side was assessed in a face-to-face interview
Affected side (part 2 only) | At baseline
  - Affected side (left or right) was assessed by the clinician
Trauma mechanism (low energy/high energy trauma or unknown) | At baseline
  - Trauma mechanism (low energy fall or other, high energy trauma, or unknown) was assessed through face-to-face interview
Additional injuries (yes or no, with specification) | At baseline
  Additional injuries were assessed in a face-to-face interview
  * Trauma mechanism (low energy fall or other, high energy trauma, or unknown)
  * Additional injuries (yes or no, with specification)
  * Fracture classification (AO type 23-A, B or C)
Fracture classification (AO type 23-A, B or C) | At baseline
  - Fracture classification (AO type 23-A, B or C) was diagnosed by the clinician
Date of scanning | At baseline
  Date of scanning was documented by the clinician
Date of brace fitting | At baseline
  Date of brace fitting was documented by the clinician.
Date of brace removal | At baseline
  Date of brace removal was documented by the clinician. If brace was removed early, it was documented how treatment was continued (in patients only).
Adherence to intervention | At baseline
  Adherence to the intervention was checked (yes/no) and reasons for not adhering were documented by the clinician

CONTACTS AND LOCATIONS:
Locations (1):
- VieCuri MC, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Janzing HMJ, Bessems SAM, Ligthart MAP, Van Lieshout EMM, Theeuwes HP, Barten DG, Verhofstad MHJ. Treatment of dorsally dislocated distal radius fractures with individualized 3D printed bracing: an exploratory study. 3D Print Med. 2020 Aug 18;6(1):22. doi: 10.1186/s41205-020-00075-4. PMID 32809083